CLINICAL TRIAL: NCT03172728
Title: Psycho-education Intervention for Postpartum Obsessive Compulsive Disorder (OCD) and it's Influence on Symptom Severity and Treatment Self Referral Rates: A Prospective Randomized Double Blinded Control Trial
Brief Title: Psycho-education Intervention for Postpartum OCD and it's Influence on Symptom Severity and Treatment Self Referral Rates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-16-GA-0658-CTIL
Record Dates: First submitted 2017-05-22; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic intervention- psycho-education pamphlet (Experimental): Psycho-education information (appendix 1) will be provided by research assistant in a pamphlet and audio recording, with a written referral to the women's mental health services in case symptoms arise. This psycho-education information will be sent again by Qualtrics 4 weeks later and women will be prompted to read it again. Women who do not respond within a week will be contacted by a research assistant and reminded to respond.
  In the end of the reading material, there will be a reading confirmation question. In the case that a participant will not answer this question or if the answer will suggest that the participant did not read the material, the research assistant will contact her by phone to confirm the reading.
  Interventions: Behavioral: psycho-education pamphlet
- Control group (No Intervention): Control group will receive general psychoeducation about the emotional after effects of childbirth in a pamphlet and audio recording and the phone number for the women's mental health services. This psychoeducation information will be sent again by Qualtrics 4 weeks later and women will be prompted to read it again. Women who do not respond will be contacted by a research assistant within a week and reminded to respond.
  In the end of the reading material, there will be a reading confirmation question. In the case that a participant will not answer this question or if the answer will suggest that the participant did not read the material, the research assistant will contact her by phone to confirm the reading.

INTERVENTIONS:
Behavioral: psycho-education pamphlet — psycho-education intervention, based on Cognitive Behavioral Therapy, that is easy to provide and feasible in standard perinatal care. It is intended to increase awareness of obsessive thoughts and to decrease anxiety and encourage treatment seeking.
  Arms: Therapeutic intervention- psycho-education pamphlet

SUMMARY:
The rationale for conducting the experiment including quantitative measures and a description of the method of recruitment:

This study provides psycho-educational intervention aimed at raising awareness of post partum Obsessive-Compulsive disorder (OCD) , reducing the intensity of symptoms and increase of self referral to treatment. Various studies report that 1-11% of women after childbirth suffer from OCD. A part of this population suffered from the disorder prior to giving birth and for some this is a first outbreak. This is a psychological disorder characterized by obsessions and compulsions. The disorder can appear or worsen at any time , and is characterized by different content depending on the stage of life. Obsessional thoughts after birth often includes harming the baby which alarms the woman and the surrounding, and affects her ability to care for the baby and develop a beneficial relationship with him. Studies support a bio-psycho-social model of OCD .and that adjustment period and physical changes after childbirth can be create a psychological biological and environmental background, to the development or worsening of OCD in women who suffer from or are prone to the disorder.

The present study deals with psycho-educational information which will be given to women after birth who were identified as susceptible to develop OCD. The information will be delivered in the maternity ward through written and recorded data , and sent through the system Qualtrics 4 weeks after birth. Psycho-education is an important first step in Cognitive Behavioral therapy for OCD and may lead to anxiety reduction and commitment to treatment. The information sent in the study is similar to the information provided at the beginning of standard Cognitive Behavioral Therapy.Women will be recruited from the maternity ward at Lis Maternity Hospital. In order to identify women at risk for OCD, All women in the maternity ward will be asked to fill a short questionnaire. Women found at risk or as suffering from OCD will be invited to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women are 48 hours after birth, meet the criteria for OCS (obsessive compulsive symptoms) or have previous history of OCD.
* Capable of filling computerized questionnaires.
* Capable of giving informed consent.

Exclusion Criteria:

* Substance use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Obsessive Compulsive Inventory-Revised questionnaire | Change from 48 hours post partum obsessive compulsive symptoms, at 8 weeks after labor.
  The Obsessive-Compulsive Inventory (OCI) was developed to help determine the severity of obsessive compulsive disorder (OCD). The OCI consists of 42 items composing 7 subscales: Washing, Checking, Doubting, Ordering, Obsessing (i.e. having obsessional thoughts), Hoarding, and Mental Neutralising. Each item is rated on a 5-point (0-4) scale of symptom distress.

IPD SHARING:
Plan to Share IPD: No